CLINICAL TRIAL: NCT03017781
Title: An Observational Longitudinal Study in Offspring of Parents With Bipolar Disorder to Evaluate the Relationship of Impairment in Psychosocial Functioning With the Manifestation of Mood Symptoms Over 24 Months
Brief Title: A Study of the Relationship of Psychosocial Function With Mood Symptoms in Offspring of Parents With Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108257; NOPRODBIP0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-12-20; First posted 2017-01-11 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; High-Risk Off-Spring; Psychosocial Functioning
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Offspring (15-25 years old) of parents with Bipolar Disorder (BD) with at least mild impairment in psychosocial functioning were observed to evaluate the relationship of impairment in psychosocial functioning with the manifestation of mood symptoms over 24 months
- Control Group: A group of offspring of bipolar parents with no impairment in psychosocial functioning will be used for comparison.

SUMMARY:
The primary purpose of this study is to compare, over 24 months, the time spent with clinically significant mood symptoms (ie, mania, depression), as measured by the Longitudinal Interval Follow-Up Evaluation (LIFE) and the Psychiatric Status Rating Scale (PSR), in offspring of bipolar parents with and without at least mild impairment in psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at least one parent who meets the criteria for diagnosis of Bipolar I disorder (BD-I) or Bipolar II disorder (BD-II), as confirmed by the Mini International Neuropsychiatric Interview (MINI) administered to the parent. MINI will be administered to parent if the history of BD is endorsed by Family Index of Risk for Mood (FIRM) or other medical information (psychiatrist, medical records). The MINI can be administered to the parent remotely through the telephone or video call if an in-person interview is not feasible due to logistical reasons. A diagnosis Bipolar Disorder Not Otherwise Specified in the parent would not qualify for eligibility
* Participants must be either drug-naive, or on stable treatment for at least 4 weeks.
* Participants (and/or their parents as applicable) must sign an Informed Consent Form (ICF) allowing data collection and source data verification in accordance with local requirements and/or sponsor policy. Adolescents (minors) who in the judgment of the investigator are capable of understanding the nature of the study can be enrolled only after obtaining consent of a legally acceptable representative. Assent must be obtained from any participating adolescents (minors), if applicable
* Participants must be willing and able to complete self-reported assessments via mobile electronic device, and to wear a wrist actigraphy device for the duration of the study

Exclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM) -IV Diagnosis of bipolar I or bipolar II disorder
* DSM-IV Diagnosis of schizophrenia, schizophreniform or schizoaffective disorder
* DSM-IV Diagnosis of neurodevelopmental disorders
* An intelligence quotient (IQ) score less than (<) 80 as determined by Kaufman Brief Intelligence Test (K-BIT)
* Uncorrected hypothyroidism or hyperthyroidism

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Offspring of parents with Bipolar Disprder (BD) will be recruited primarily at selected sites which are already conducting research in prodromal BD and have the necessary setup and resources already in place to conduct such a study.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Weeks Spent With Clinically Significant Mood Symptoms in a 24-Month Longitudinal Study Period, Which will be Derived From the Longitudinal Interval Follow-up Evaluation (LIFE) | Up to 24 months
  The LIFE is a semi-structured interview developed for prospectively following the course of psychiatric disorders; the LIFE collects detailed psychosocial, psychopathologic and treatment information for a 6-month follow-up interval.
Proportion of Weeks Spent With Clinically Significant Mood Symptoms in a 24-Month Longitudinal Study Period, Which will be Derived From the Psychiatric Status Rating (PSR) | Up to 24 months
  Weekly symptomatic status, including symptom severity, will be assessed through the Psychiatric Status Ratings (PSRs). Ratings of 1 or 2 on the PSR represent remission or minimal symptoms; ratings of 3 or 4 represent clinically significant subthreshold symptoms; a rating of 5 represents a current episode of hypomania or moderate major depression; and a rating of 6 represents a current episode of mania or severe depression.

SECONDARY OUTCOMES:
Global Assessment of Functioning (GAF) | Up to 24 months
  GAF is a numeric scale (1 through 100) used by mental health clinicians and physicians to rate the social, occupational, and psychological functioning of adults.
Bipolar Prodrome Symptom Interview and Scale-Prospective (BPSS-P) | Up to 24 months
  The BPSS-P assesses the onset and severity of prodromal symptoms and is divided into 3 sections: Mania, Depression, and General Symptom Index. The BPSS-P yields a total score, and separate scores each of the 3 sections.
Mini International Neuropsychiatric Interview (MINI) | Up to 24 months
  MINI is a short, structured diagnostic interview for psychiatric disorders, divided into modules identified by letters, each corresponding to a diagnostic category.
Neuropsychological Testing | Up to 24 months
  Neuropsychological testing will be performed using a computerized test battery, as well as "paper-based" neuropsychological tasks to have a better understanding of the contribution of cognitive function and potential deficits in domains relevant for Bipolar Disorder (BD) to the clinical symptoms and longitudinal trajectory over 24 months.
General Behavioral Inventory (GBI) | Up to 24 months
  GBI is a 73-item, self-assessment questionnaire designed to assess symptoms of depression and mania/hypomania (18 or higher for depression or 13 or lower for mania/hypomania).
Changes in Quality of Life as Assessed Using the Qol (EQ-5D-5L) Scale | Up to 24 months
  EQ-5D-5L is a quality of life (QoL) preference-based measure of health outcome that provides a simple descriptive profile and a single index value for health status. The instrument consists of 5 dimensions of health, each with 5 levels of problems.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (20):
- United States (20):
  - Culver City, California
  - Lemon Grove, California
  - Los Angeles, California
  - Palo Alto, California
  - Panorama City, California
  - Tampa, Florida
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Glen Oaks, New York
  - Rochester, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Austin, Texas
  - Dallas, Texas
  - El Paso, Texas

REFERENCES:
- [Derived] Pandina G, DelBello MP, Rassnick S, Solanki B, Canuso CM, Fristad MA, Correll CU, Nurnberger JI Jr, Singh MK, McInnis MG, Atkinson S, Stedman M, Goes FS, Strakowski SM, Greer TL, Nierenberg AA, Salvadore G, Drevets WC. Clinical outcomes of youth at familial risk for bipolar disorder: A 2-year longitudinal, observational study. J Affect Disord. 2026 Jan 15;393(Pt B):120492. doi: 10.1016/j.jad.2025.120492. Epub 2025 Oct 15. PMID 41106637